CLINICAL TRIAL: NCT07322705
Title: Can Perineal Post-Free Traction in Hip Arthroscopy Effectively Reduce Perineal Complications? A Multicenter Prospective Randomized Controlled Trial
Brief Title: Can Perineal Post-Free Traction in Hip Arthroscopy Effectively Reduce Perineal Complications?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ChunBao Li (Other)
Responsible Party: Sponsor-Investigator, ChunBao Li, Director of the Department of Sports Medicine, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024KY0158-KS001
Record Dates: First submitted 2025-11-17; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Femoroacetabular Impingement Syndrome
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perineal Post-Free Traction (Experimental)
  Interventions: Procedure: Perineal Post-Free Traction
- Perineal Post Traction (Active Comparator)
  Interventions: Procedure: Perineal Post Traction

INTERVENTIONS:
Procedure: Perineal Post-Free Traction — Traction achieved with a thoraco-abdominal belt and contralateral groin strap; operating table tilted 10-15° Trendelenburg; gradual 10-20 kg distraction under fluoroscopy to 8-10 mm joint space. No perineal post is used, eliminating direct perineal pressure.
  Arms: Perineal Post-Free Traction
Procedure: Perineal Post Traction — Standard traction table with padded perineal post placed against the groin providing counter-traction; affected limb distracted under fluoroscopy to 8-10 mm joint space while contralateral limb is abducted.
  Arms: Perineal Post Traction

SUMMARY:
The goal of this clinical trial is to analyze the impact of perineal post-free traction versus traditional perineal post traction on perineal complications in hip arthroscopy. The main question it aims to answer is:

• Can Perineal Post-Free Traction in Hip Arthroscopy Effectively Reduce Perineal Complications? Researchers will compare the perineal-post-free traction group with the conventional perineal-post traction group to see if the former decreases perineal complications and improves efficiency without compromising surgical outcomes.

Participants will:

* Undergo either perineal-post-free or standard perineal-post traction during hip arthroscopy
* Complete nerve-injury checks on day 1 and at discharge, and hip-function questionnaires (VAS, mHHS, IHOT-12, HOS) at 3 months
* Allow collection of operating times, hospital stay, and direct medical costs for economic analysis

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 to 60 years;
* Met the diagnostic criteria of femoroacetabular impingement syndrome (FAI) and indicated for hip arthroscopy based on patient history, symptoms, signs, physical examination, imaging (pelvic anteroposterior view, frog-leg view, CT 3D reconstruction, MRI), and diagnostic injections;
* Able to read and sign the informed consent form.

Exclusion Criteria:

* History of high-energy hip trauma, previous ipsilateral or contralateral hip surgery, avascular necrosis of the femoral head, slipped capital femoral epiphysis, Perthes disease, severe osteoporosis, tumors, acetabular stress fractures, or proliferative or immune hip diseases;
* Diseases causing groin numbness, foot numbness, sexual dysfunction, urinary dysfunction, skin injuries, perineal injuries, nerve injuries, radicular pain, inner or outer thigh numbness;
* Abnormal heart, lung, liver, kidney function, severe coagulation disorders, poorly controlled diabetes, judged by the researcher to have an infection risk;
* Consciousness disorders, psychiatric disorders, or neuromuscular dysfunction affecting lower limb function;
* Active infection foci (systemic or local infectious lesions);
* Pregnancy, lactation, or planned pregnancy during the clinical study period;
* Participation in another clinical trial within the past 3 months;
* Patients deemed unsuitable for the clinical trial by the researcher for other reasons.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 270 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of perineal nerve injury | The first day after surgery
  The incidence of perineal nerve injury included: perineal numbness, pain, soft tissue injury, sexual function and urinary dysfunction.sexual function and urinary dysfunction.

SECONDARY OUTCOMES:
The incidence of pain, numbness, soft tissue injury in other places | The first day after surgery
  Lower limb ankle numbness and soft tissue injury; the contralateral groin pain, numbness and soft tissue injury; chest pain, numbness, soft tissue injury with fixed place
Patients at discharge perineum area incidence of nerve injury | 7 days after surgery
  Patients at discharge perineum area incidence of nerve injury include: perineum area numbness, pain, soft tissue injuries, sexual and urinary dysfunction.
Intraoperative traction time | During surgery (intraoperatively)
  Intraoperative traction time
Preoperative preparation time | Immediately before surgery (preoperatively)
  Preoperative preparation time
Operating time | During surgery (intraoperatively)
  Operating time
The average length of hospital stay after surgery | 6 weeks after surgery
  The average length of hospital stay after surgery
Postoperative joint function assessment | 3 months after surgery
  Visual Analog Scale (VAS) (range 0-10; higher scores indicate worse outcomes).
Postoperative joint function assessment | 3 months after surgery
  Modified Harris Hip Score (mHHS) (range 0-100; higher scores indicate better outcomes).
Postoperative joint function assessment | 3 months after surgery
  Hip Outcome Score (HOS) (range 0%-100%; higher scores indicate better outcomes).
Economic Evaluation - Pain Intensity | 14 days after surgery
  This study will conduct an economic evaluation from a healthcare sector and societal perspective. Pain intensity is assessed using the Visual Analog Scale (VAS), a unidimensional measure reported as scores on a 0-100 mm scale. Effectiveness analysis will incorporate this clinical outcome. Safety will be evaluated by monitoring the incidence of adverse events within 3 months postoperatively.
Economic Evaluation - Hip Function | 14 days after surgery
  This study will conduct an economic evaluation from a healthcare sector and societal perspective. Hip function is assessed using the modified Harris Hip Score (mHHS), a measure specifically for hip dysfunction and related symptoms, reported as scores on a 0-100 scale. Effectiveness analysis will incorporate this clinical outcome. Safety will be evaluated by monitoring the incidence of adverse events within 3 months postoperatively.
Mean Total Healthcare Cost per Patient within 14 Days Postoperatively | Data collection period: From randomization until 14 days postoperatively.
  This is the cost input measure for the economic evaluation, adopting a healthcare system perspective. All direct medical costs related to the surgery and subsequent care from the day of surgery until 14 days postoperatively will be collected via the Hospital Information System. Costs include fees for surgery, anesthesia, medical supplies, hospitalization, medication, imaging and laboratory tests, and additional costs for managing complications. The mean total cost per patient (in Chinese Yuan, CNY) will be calculated separately for the "conventional perineal-post traction group" and the "perineal-post-free traction group".